CLINICAL TRIAL: NCT06816498
Title: An Open-label, Single-center, Single-participant Study of an Experimental Antisense Oligonucleotide Treatment for a Patient With LMNB1 Mutation Associated Autosomal Dominant Leukodystrophy (ADLD)
Brief Title: Personalized Antisense Oligonucleotide Therapy for A Single Participant With LMNB1 Mutation Associated Autosomal Dominant Leukodystrophy (ADLD)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-011942
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Autosomal Dominant Leukodystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-LMNB1-001

INTERVENTIONS:
Drug: nL-LMNB1-001 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with Autosomal Dominant Leukodystrophy (ADLD) due to LMNB1 mutation

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with Autosomal Dominant Leukodystrophy (ADLD) due to LMNB1 mutation

ELIGIBILITY:
Inclusion Criteria:

* Informed consent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s).
* Autosomal dominant adult-onset leukodystrophy (ADLD) caused by an LMNB1 duplication mutation
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records.
* Willingness to follow contraceptive guidance during the intervention period and for at least 40 weeks after the last dose of study intervention

Exclusion Criteria:

* Participant has any condition that in the opinion of the Site Investigator, would ultimately prevent the completion of study procedures

Ages: 51 Years to 51 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Gait | Baseline to 24 months
  Change in gait from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration as measured by gait motion analysis
Gait | Baseline to 24 months
  Change in gait from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration as measured by 6-minute walk test
Gait | Baseline to 24 months
  Change in gait from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration as measured by 25-feet walk test
Neurological functioning | Baseline to 24 months
  Change in neurological functioning results from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration as measured by formal neuro-psychological evaluation (abnormalities in cognitive functioning such as memory, visual function, and language function).
Brain atrophy | Baseline to 24 months
  Change in degree of brain atrophy from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration as measured by brain MRI

SECONDARY OUTCOMES:
Urodynamics | Baseline to 24 months
  Change from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration in urodynamic study (normal or abnormal bladder activity).
Autonomic function | Baseline to 24 months
  Change from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration in autonomic function as measured by % anhidrosis from thermoregulatory sweat test
Autonomic function | Baseline to 24 months
  Change from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration in autonomic function as measured by Quantitative Axon Reflex Sweat Test sweat output (uL)
Autonomic function | Baseline to 24 months
  Change from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration in autonomic function as measured by supine and standing catecholamines levels
Autonomic function | Baseline to 24 months
  Change from baseline at 6-, 12-, 18- and 24-months post nL-LMNB1-001 administration in autonomic function as measured by 24-hour ambulatory blood pressure monitoring
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Baseline to 24 months
Incidence of Treatment-Emergent abnormalities in physical and neurological exams [Safety and Tolerability] | Baseline to 24 months
Incidence of Treatment-Emergent abnormalities in safety labs (CSF, chemistry, hematology, coagulation, and urinalysis) [Safety and Tolerability] | Baseline to 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided